CLINICAL TRIAL: NCT02571725
Title: A Phase 1-2 Study of the Combination of Olaparib and Tremelimumab, in BRCA1 and BRCA2 Mutation Carriers With Recurrent Ovarian Cancer
Brief Title: PARP-inhibition and CTLA-4 Blockade in BRCA-deficient Ovarian Cancer
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: New Mexico Cancer Research Alliance (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INST 1419
Record Dates: First submitted 2015-10-06; First posted 2015-10-08 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Neoplasms
Keywords: Ovarian cancer; Fallopian tube cancer; Peritoneal cancer; PARP; BRCA; Immunotherapy; Olaparib; Tremelimumab; CTLA4
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Peritoneal Neoplasms | interventions — olaparib; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Olaparib and Tremelimumab (Experimental): Each cycle is 28 days:
  Olaparib at 300 mg, orally, twice daily + Tremelimumab at 10 mg/kg, intravenously, every 4 weeks for the first 6 doses, then every 12 weeks until disease progression or unacceptable toxicity.
  * If 1 of the first 3 patients experiences a regimen-limiting toxicity (RLT), 3 more patients will be treated with 10 mg/kg Tremelimumab in Phase 1. If 2 or more of 6 patients experience RLT, then 6 mg/kg Tremelimumab will be tested
  * If at 6 mg/kg, 1 or more of 3 patients experience RLT, 3 patients will be treated at 3 mg/kg Tremelimumab
  * If at 3 mg/kg, 1 or more patients experience RLT, the study will be discontinued for safety purposes
  In Phase 2, patients will receive doses of Olaparib and Tremelimumab determined in the Phase 1 portion as described above, based on tolerability.
  Interventions: Drug: Olaparib; Drug: Tremelimumab

INTERVENTIONS:
Drug: Olaparib — Olaparib starts concomitantly with the first dose of Tremelimumab
  Other Names: AZD-2281; Lynparza
Drug: Tremelimumab — 3 to 6 patients will be treated at 10 mg/kg depending on RLT observed in the first 3 patients. If 0 out of 3 or 1 out of 6 patients experienced a RLT at 10 mg/kg, then this dose will be considered at the recommended phase 2 dose (RP2D). If 2 out of 6 patients experience RLT at this dose within 56 days, then dose reductions as detailed in the Arm description will be carried out.
  Other Names: CP-675,206

SUMMARY:
Of the approximately 21,000 cases of ovarian cancer diagnosed annually in the U.S, ten percent are attributed to hereditary syndromes, most commonly the result of mutations in the breast cancer susceptibility genes 1 or 2 (BRCA1 or BRCA2). Mutation in these genes results in the inability to repair double-stranded breaks in DNA. Treating these tumors with poly(adenosine diphosphate [ADP]-ribose) polymerase (PARP) inhibitors results in the specific killing of BRCA negative cells by blocking a second DNA-repair mechanism. Treatment of ovarian cancer patients with PARP inhibitors has resulted in improved progression free survival (PFS), but not overall survival (OS). It's not completely understood why this is the case, but some preclinical studies using ovarian cancer models in mice have suggested that combining PARP inhibitors with immune system modulators like T cell checkpoint inhibitors improves long-term survival.

Therefore, the purpose of this study is to evaluate the safety and efficacy of a combination of a PARP inhibitor (Olaparib) with a T cell checkpoint inhibitor (the anti-CTLA-4 antibody Tremelimumab) in women with recurrent BRCA mutation-associated ovarian cancer.

DETAILED DESCRIPTION:
The mechanism of action of Olaparib, a potent inhibitor of mammalian PARP-1, PARP-2, and PARP-3, has been proposed to involve the trapping of inactivated PARP onto single-stranded breaks preventing their repair and generating a potential block for cellular DNA replication. In tumors with homologous recombination deficiency, such as those with BRCA mutations, single agent treatment with Olaparib can lead to cell death and tumor regressions by a process known as synthetic lethality.

Tremelimumab is a human monoclonal immunoglobulin G2 (IgG2) antibody specific for human cytotoxic T lymphocyte-associated antigen 4 (CTLA-4), a co-inhibitory receptor expressed on activated T cells. Tremelimumab has been shown to block the inhibitory signal mediated by interaction of human CTLA-4 on activated T cells with B7-1 and B7-2 on antigen-presenting cells. This is thought to maintain T cell activation in the tumor microenvironment and promote the establishment of tumor-specific immune responses.

Like melanoma, ovarian cancer is associated with significant tumor heterogeneity, and is also a rational target for immune therapy. Although antitumor effects have been observed in patients with epithelial ovarian cancer in response to anti-CTLA-4 antibody treatment, evidence of clinical disease regression has not been demonstrated. Based on data indicating that a subset of ovarian cancers associated with germline mutations in BRCA1/2 genes may be more immunogenic, we hypothesized that BRCA-negative tumors would be particularly vulnerable to checkpoint blockade, and that immune priming with targeted cytotoxic therapy using a PARP-inhibitor would sensitize ovarian tumors to immune therapy and optimize patient survival. We have demonstrated this in pre-clinical models of high grade BRCA1-negative ovarian cancer.

Based on significant therapeutic benefit demonstrated in pre-clinical models, this clinical trial evaluates the combination of Olaparib and Tremelimumab in women with recurrent BRCA-deficient ovarian cancers.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma for which standard curative measures do not exist.
* Patients must have a confirmed germline mutation in the BRCA1 or BRCA2 gene
* Patients must have measurable disease as defined by World Health Organization (WHO) criteria: at least 1 lesion that can be accurately measured in at least 1 dimension (longest diameter to be recorded). Each lesion must be >1.0cm when measured by CT, MRI, or caliper measurement by clinical exam; or >2.0cm when measured by chest x-ray. Lymph nodes must be >1.5cm in short axis when measured by CT or MRI
* Patients with platinum-sensitive or platinum-resistant disease are eligible
* Patients must have received at least 1 prior course of platinum-based chemotherapy for the management of primary disease including carboplatin, cisplatin, or another platinum compound
* There are no restrictions on the total number of prior regimens patients may have received
* Gynecologic Oncology Group (GOG) performance status of 0, 1, or 2
* Adequate organ and marrow function as defined below:

  * Absolute neutrophil count (ANC) >1,500/mcl
  * Platelets > 100,000/mcl
  * Creatinine < 1.5x the institutional upper limit of normal (ULN)
  * Bilirubin < 1.5x ULN
  * Aspartate aminotransferase and Alanine aminotransferase < 3x ULN
  * Alkaline phosphatase < 2.5x ULN
* Women of child-bearing potential must have a negative pregnancy test prior to study entry and agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 180 days following completion of therapy
* Ability to understand and the willingness to sign a written informed consent document
* Patients must meet pre-entry requirements as specified

Exclusion Criteria:

* Recovery from effects of recent surgery, radiotherapy, or chemotherapy must be demonstrated
* Patients should be free of active infection requiring antibiotic therapy (except for uncomplicated urinary tract infections)
* Hormonal therapy directed at treatment for the cancer must be discontinued at least 1 week prior to enrollment. Hormone replacement therapy for symptom management is permitted.
* Any other therapy directed at treating the cancer including chemotherapy, biologic/targeted agents, and immunologic agents, must be discontinued at least 3 weeks prior to enrollment.
* Any prior radiation therapy must be discontinued at least 4 weeks prior to enrollment.
* A history of autoimmune disorders other than vitiligo (e.g., psoriasis, extensive atopic dermatitis, asthma, inflammatory bowel disease, multiple sclerosis, uveitis, vasculitis), chronic inflammatory condition, or any condition requiring concurrent use of any systemic immunosuppressants or steroids for any reason are excluded from the study. Any patient with an allo-transplant of any kind would be excluded as well, including xenograft heart valve. Mild, intermittent asthma requiring only occasional beta-agonist inhaler use or mild localized eczema will not be excluded.
* Chronic use of immune-suppressive drugs (i.e., systemic corticosteroids used in the management of cancer or non-cancer related illnesses, e.g., COPD).
* Known HIV-positive patients and those with other acquired/inherited immunodeficiencies are ineligible due the possibility of affecting the response to tremelimumab, and the higher risk of active opportunistic infections.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to olaparib or tremelimumab, or other agents used in study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Concomitant use of known potent cytochrome P450 isoform 3A4 (CYP3A4) inhibitors
* Persistent toxicities (> Common Terminology Criteria for Adverse Event (CTCAE) grade 2) caused by prior cancer therapy, excluding alopecia
* Must not be pregnant or nursing as the potential of this regimen to harm nursing infants has not been evaluated.
* Patients who are receiving any other investigational agent

For Phase 2, the inclusion/exclusion criteria above apply. In addition, the following exclusion criteria apply:

* Resting electrocardiogram with corrected QT interval (QTc) >470msec on two or more time points within a 24hr period, or a family history of long QT syndrome
* Patients who have previously received anti-CTLA-4 antibody therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-02-23 (Actual); Primary Completion 2020-12-02 (Actual); Study Completion 2027-07-15 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Recommended Phase 2 Dose (RP2D) | Within 56 days of first treatment (up to 2 years)
  The RP2D will be based on determination of the regimen-limiting toxicity (RLT), i.e., toxicity induced by the immunological agent that limits the administration of the backbone therapy (Olaparib).
  RLT is defined as the following toxicities occurring during the first two cycles (56 days) of treatment (with the combination of Olaparib and Tremelimumab):
  * Any grade 4 non-hematological toxicity that is treatment-related with the exception of alopecia, nausea and vomiting or lymphopenia.
  * Any grade 3 non hematological toxicity that is treatment related that results in delay of Olaparib by greater than 4 weeks.
  * Delay in starting the second cycle by more than 2 weeks due to toxicity attributable to Tremelimumab.
  The RP2D of Tremelimumab is one that does not induce RLT in more than 1 of 6 patients.
Phase 2: Objective response rate (ORR) | 2 years
  Patients will be followed both clinically and radiographically every 12 weeks. Responses will be assessed using immune-related response criteria (irRC) (Wolchock et al 2009) in which tumor volume measurements are assessed along with the emergence of new measurable lesions. Each net percentage change in tumor burden accounts for the size and growth kinetics of both old and new lesions as they appear. The sum of the product of the diameters for all index lesions identified prior to enrollment is the immune-related sum of products of diameters (irSPD). Complete Response (CR), Disappearance of all tumor lesions; Partial Response (PR), >=50% decrease relative to the baseline irSPD. ORR = proportion of patients whose best overall response is either CR or PR.

SECONDARY OUTCOMES:
Phase 2: Progression free survival (PFS) | 5 years
  PFS is defined as the time between the first dose of study therapy and the earliest of progression or death. Patients will be followed both clinically and radiographically every 12 weeks. Responses will be assessed using immune-related response criteria (irRC) (Wolchock et al 2009) in which tumor volume measurements are assessed along with the emergence of new measurable lesions. Each net percentage change in tumor burden accounts for the size and growth kinetics of both old and new lesions as they appear. The sum of the product of the diameters for all index lesions identified prior to enrollment is the immune-related sum of products of diameters (irSPD). New lesions alone do not qualify as progressive disease. Progressive disease is >= 25% increase in the irSPD (based on irSPD of all index lesions and any measurable new lesions) over the nadir irSPD, or the occurrence of any new measurable lesions if the SPD nadir is "0."

CONTACTS AND LOCATIONS:
Overall Officials: Sarah F Adams, MD, Principal Investigator — University of New Mexico Comprehensive Cancer Center
Locations (5):
- United States (5):
  - Moffitt Cancer Center, Tampa, Florida
  - Southwest Gynecologic Oncology Associates, Albuquerque, New Mexico
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - The Ohio State University, Columbus, Ohio
  - University of Virginia Cancer Center, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of New Mexico Comprehensive Cancer Center — http://cancer.unm.edu/
- See also: New Mexico Cancer Care Alliance — http://nmcca.org/